CLINICAL TRIAL: NCT01494844
Title: Comfort Evaluation of Non-Invasive Respiratory Monitor Interfaces
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Oridion (Industry)
Responsible Party: Principal Investigator, Jonathan B. Waugh, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: X110421003; 413525 (Other Grant/Funding Number: Oridion Capnography Inc.)
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Respiratory Device Comfort
Keywords: Patient Monitoring; Capnography; Human Engineering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device interface comfort assessment (Other): Single group rates one noninvasive respiratory monitoring interface and then another.
  Interventions: Device: Respiratory monitor patient interface.

INTERVENTIONS:
Device: Respiratory monitor patient interface. — Wear each interface for 20 minutes
  Other Names: Masimo Rainbow Acoustic Monitoring sensor; Oridion Smart Capnoline Plus H sensor

SUMMARY:
This research study will test the comfort of two noninvasive respiratory monitoring sensors (the connection to a monitor worn by a person-not the monitor). The two sensors, Masimo Rainbow Acoustic Monitoring sensor and Oridion Smart Capnoline Plus H sensor, are cleared by the U.S. Food and Drug Administration (FDA) and currently used in the clinical setting. People who enter into the study will wear the two interfaces, one after the other, for 20 minutes each (10 minutes with a small flow of air to the nostrils and 10 minutes without) and rate the comfort of each with a seven question survey. A total of 30 participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Normal body temperature
* Between the ages of 19-65 years
* Self-report as feeling to be in typical health
* No skin irritation face or neck where a sensor would be placed.
* School of Health Professions student

Exclusion Criteria:

* Any injury or condition that would affect assessment of comfort.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Comfort Rating Self-Report Instrument | 5 Minutes
  A seven-question written instrument constructed in the style of descriptive analogue to evaluate multiple facets of device comfort. Answer choices allow either ordinal ranking (one requires a ranking on a continuous time scale).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Waugh, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Waugh JB, Epps CA. Comfort evaluation of noninvasive respiratory monitoring interfaces. Respir Care 2011; 56(10): 1722.